CLINICAL TRIAL: NCT05320107
Title: Unraveling the Aesthetic Mind in Anhedonia, Insights From Pharmacological Imaging of the Human Brain: A Single-blind, Randomized, Placebo-controlled Cross-over Study
Brief Title: The Effect of Ketamine on Aesthetics and Role for Antidepressant Effects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Principle Investigator, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PSY-NIL-0010
Record Dates: First submitted 2022-02-26; First posted 2022-04-11 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine first, then placebo (Experimental): 0.5mg/kg bodyweight (or 0.25mg/kg bodyweight) ketamine, will be determined in pilot study, then placebo
  Interventions: Drug: Ketamine; Drug: Placebo
- Placebo frist, then ketamine (Experimental): 0.9% NaCl, then ketamine
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — 0.5mg/kg bodyweight (or 0.25mg/kg bodyweight) ketamine, will be determined in pilot study
Drug: Placebo — 0.9% NaCl

SUMMARY:
The aim of this study is to assess the impact of ketamine on aesthetic perception and processing. This study assesses the role of these effects in facilitating ketamine's antidepressant properties, with a focus on anhedonia. To address this aim, 25 patients with major depressive disorder and 35 healthy controls will be assessed twice with magnetic resonance imaging, once after administration of intravenous ketamine (subanesthetic dose) and once after administration of placebo.This study has a single-center, placebo-controlled, cross-over study design. During MRI, structural, resting state, and functional imaging will be performed. Functional imaging will comprise aesthetic processing, reward, and sexual arousal paradigms. In addition, various neuropsychological scales assessing depressive symptoms, anhedonia, and aesthetic processing will be performed. Eligibility for participation will be assessed during a screening visit, a follow up visit will end study participation.

ELIGIBILITY:
Inclusion Criteria:

* General health based on medical history and physical examination
* Psychiatric health based on structured clinical interview for DSM-5 (SCID) for healthy controls
* Major depressive episode (first or recurrent) based on structured clinical interview for DSM-5 and ICD-10 for patients
* Age 18 to 55 years
* Right-handedness (due to potential lateralization effects of lefthanded subjects)
* Willingness and competence to sign the informed consent form

Exclusion Criteria:

* Current or history of neurological disease
* Current medical illness requiring treatment
* Psychiatric diagnosis for healthy individuals
* Psychiatric comorbidity with the exception of anxiety disorders for depressed individuals
* Pregnancy or current breastfeeding
* Current or former substance abuse
* Previous ketamine use in lifetime
* Any contraindication for MRI (e.g., MR incompatible implants, etc.) including dental implants causing signal artifacts
* Failure to comply with the study protocol or to follow the instruction of the investigating team

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
BOLD signal assessed with fMRI during aesthetic paradigm | Change from baseline to up to 4 weeks
  Difference in Blood Oxygen Level Dependent (BOLD) signal assessed with functional magnetic resonance imaging (fMRI) between ketamine and placebo condition during an aesthetic processing task
BOLD signal assessed with fMRI during reward paradigm | Change from baseline to up to 4 weeks
  Difference in Blood Oxygen Level Dependent (BOLD) signal assessed with functional magnetic resonance imaging (fMRI) between ketamine and placebo condition during a reward processing task
BOLD signal assessed with fMRI during sexual arousal paradigm | Change from baseline to up to 4 weeks
  Difference in Blood Oxygen Level Dependent (BOLD) signal assessed with functional magnetic resonance imaging (fMRI) between ketamine and placebo condition during a sexual arousal paradigm
Levels of pleasantness assessed during aesthetic fMRI task | Change from baseline to up to 4 weeks
  Level of pleasantness (Numbered scale) of aesthetic stimuli during aesthetic paradigm task
Number of of chills assessed during aesthetic fMRI task | Change from baseline to up to 4 weeks
  Number of chills in response to aesthetic stimuli during aesthetic paradigm task
BOLD signal assessed with fMRI during resting state | Change from baseline to up to 4 weeks
  Difference in Blood Oxygen Level Dependent (BOLD) signal assessed with functional magnetic resonance imaging (fMRI) between ketamine and placebo condition during resting state

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria